CLINICAL TRIAL: NCT04175236
Title: Analysis of a Short Assessment of Post Intensive Care Syndrome (PICS)
Status: Completed | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: PICS
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Postintensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To present a proposal for a set of outcome measurement instruments (OMIs) of post intensive care syndrome (PICS) in settings of outpatient healthcare service.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, whose intensive care treatment has already been completed

  * The patients were interviewed in the Klinikum Ernst von Bergmann, Peumologisches Beatmungszentrum, Bad Belzig, as well as in the pain clinic of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin

Exclusion Criteria:

Patients with a legal guardian or authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patienten aged ≥ 18 years, whose intensive care treatment has already been completed from the Klinikum Ernst von Bergmann, Peumologisches Beatmungszentrum, Bad Belzig, as well as from the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Post Intensive Care Syndrome (PICS) | 06/2018 - 11/2019
  The composite outcome measure "PICS" of the patient is measured according to Needham et al 2012: new impairment or worsening of health after intensive care unit stay and at the same time clinically significant distress in at least one of the following outcome measurement instruments: Patient Health Questionnaires (PHQ-9, PHQ-8, PHQ-4), Generalized Anxiety Disorder Scale-7 (GAD-7), Impact of Event Scale (IES), Impact of Event Scale Revised (IES-R), MiniCog, Animal Naming Test, Trail Making Test (TMT-A, TMT-B), Repeatable Battery for the Assessment of Neuropsychological Satus (RBANS), Timed Up-and-Go (TUG), Handgrip Strength, 2-Minute Walk Test (2-MWT), Short Physical Performance Battery (SPPB).

SECONDARY OUTCOMES:
Subjective Health I | 06/2018 - 11/2019
  Patients were asked to rate their quality of life, measured by EQ-5D-3L
Subjective Health II | 06/2018 - 11/2019
  Patients were asked to rate their quality of life, measured by EQ-5D-5L
Subjective Health III | 06/2018 - 11/2019
  Patients were asked to rate their quality of life, measured by WHO Disability Assessment Schedule (WHODAS 2.0)
Mental Health | 06/2018 - 11/2019
  Mental health of the patient is measured by the sum scores of the following outcome measurement instruments: Patient Health Questionnaire (PHQ-9, PHQ-8, PHQ-4), Generalized Anxiety Disorder Scale-7 (GAD-7), Impact of Event Scale (IES), Impact of Event Scale Revised (IES-R).
Cognition | 06/2018 - 11/2019
  Cognition is measured by the sum scores of the following outcome measurement instruments: MiniCog, Animal Naming Test, Trail Making Test (TMT-A, TMT-B), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Physical Health | 06/2018 - 11/2019
  Physical health is measured by the sum scores of the following outcome measurement instruments: Timed Up-and-Go (TUG), Handgrip Strength, 2-Minute Walk Test (2-MWT), Short Physical Performance Battery (SPPB).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Klinikum Ernst von Bergmann, Peumologisches Beatmungszentrum, Bad Belzig
  - Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Berlin

REFERENCES:
- [Derived] Spies CD, Krampe H, Paul N, Denke C, Kiselev J, Piper SK, Kruppa J, Grunow JJ, Steinecke K, Gulmez T, Scholtz K, Rosseau S, Hartog C, Busse R, Caumanns J, Marschall U, Gersch M, Apfelbacher C, Weber-Carstens S, Weiss B. Instruments to measure outcomes of post-intensive care syndrome in outpatient care settings - Results of an expert consensus and feasibility field test. J Intensive Care Soc. 2021 May;22(2):159-174. doi: 10.1177/1751143720923597. Epub 2020 May 14. PMID 34025756